CLINICAL TRIAL: NCT06286228
Title: Registry of Haploidentical Hematopoietic Stem Cell Transplantation in Adult With Hematologic Disease
Acronym: Haplo
Status: Not yet recruiting | Type: Observational
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Chutima Kunacheewa, lecturer, Siriraj Hospital
Other Study IDs: 751/2563(IRB4)
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Multiple Myeloma
Keywords: haploidentical hematopoietic stem cell transplantation (haploHSCT); registry
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to register hematologic patients with haploidentical hematopoietic stem cell transplantation (haploHSCT). The main questions it aims to answer are:

* 1-year progression free survival rate
* 1-year overall survival rate
* Graft-versus-host free relapsed free survival at 30-day, 100-day, 180-day and 1-year
* Chronic Graft-versus-host free relapsed free survival at 180-day and 1-year
* Rate of Neutrophil and platelet engraftment
* Efficacy of donor specific antibody desensitization
* Relapsed rate
* Primary and late graft failure
* Safety and complication of haploHSCT
* Complication of viral, bacterial, and fungal infection
* Viral reactivation
* Comparison outcomes between matched sibling donor (MSD) HSCT and matched unrelated donor (MUD) HSCT
* Comparison cost-effectiveness of treatment between matched sibling donor (MSD) HSCT and matched unrelated donor (MUD) HSCT Participants will be collected the data of baseline diagnosis, treatment, treatment results of all admission and follow-up visits from hospital medical record.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hematologic diseases indicated for treatment with haploidentical hematopoietic stem cell transplantation including

  1. Myeloid diseases (acute myeloblastic leukemia, myelodysplastic syndrome, chronic myelocytic leukemia, classical and non-classical myeloproliferative disorders)
  2. Lymphoid disease (acute lymphoblastic leukemia, lymphoma)
  3. severe aplastic anemia
* Unable to find a matched sibling donor (MSD) or matched unrelated donor (MUD), and no alternative treatments
* Eastern Cooperative Oncology Group (ECOG) 0-2
* normal AST and ALT, creatinine <2g/dL, and left ventricular ejection fraction ≥50%
* age >18 years
* Capable of informed consent and provision of written informed consent before any study procedures
* Capable of attending all study visits according to the study schedule
* Female subjects who is childbearing potential must have a negative result for pregnancy test

Exclusion Criteria:

* HIV infection, active hepatitis B, active hepatitis C
* active infection
* history of other malignancy except basal cell carcinoma and carcinoma of the cervix in situ
* A pregnant woman and/or refusal of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hematologic patients with haploidentical hematopoietic stem cell transplantation
Sampling Method: Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2029-04-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
register hematologic patients with haploidentical hematopoietic stem cell transplantation | 5 years

SECONDARY OUTCOMES:
progression free survival rate | 1 year
overall survival rate | 1 year
Chronic Graft-versus-host free relapsed free survival | at 180-day and 1-year
Relapsed rate | 5 years
Primary and late graft failure | 5 years
Rate of Neutrophil and platelet engraftment | during admission
Efficacy of donor specific antibody desensitization | during admission
Safety and complication of haploHSCT | 5 years
Complication of viral, bacterial, and fungal infection | during admission
Viral reactivation | during admission
outcomes between matched sibling donor (MSD) HSCT and matched unrelated donor (MUD) HSCT | 5 years
cost-effectiveness of treatment between matched sibling donor (MSD) HSCT and matched unrelated donor (MUD) HSCT | 5 years

IPD SHARING:
Plan to Share IPD: Undecided
Need a consensus from colleagues